CLINICAL TRIAL: NCT03642119
Title: Validation of an Objective Instrument to Measure Hot Flashes During Menopause
Acronym: FLAME
Status: Terminated | Type: Observational
Why Stopped: PI left the intuition
Sponsor: Pennington Biomedical Research Center (Other)
Responsible Party: Sponsor
Other Study IDs: PBRC 2018-027
Record Dates: First submitted 2018-08-09; First posted 2018-08-22 (Actual); Last update posted 2023-02-02 (Actual); Status verified 2022-09

CONDITIONS: Menopause; Hot Flashes
MeSH Terms: conditions — Hot Flashes

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- iButton® Validation in Perimenopause: Women in the late phase of perimenopause (based on the STRAW+10 criteria).
  Interventions: Device: iButton®

INTERVENTIONS:
Device: iButton® — Women with frequently reported hot flashes will be undergo both real world (ambulatory; field tests) and controlled (laboratory) assessments to validate the iButton® as an objective method to assess hot flash dynamics and incidence.

SUMMARY:
The overarching aim of this study is to assess the validity of the iButton®, a dual temperature and humidity sensing device (DS1923; Maxim IntegratedTM), as an objective method to assess hot flash incidence and dynamics in both a real world (ambulatory) and controlled (laboratory) setting. This study will test the overarching hypothesis that both self-report hot flashes in both an ambulatory and laboratory setting will correlate (confirm) the temperature and humidity sensing observed via the iButton® technology.

DETAILED DESCRIPTION:
Using iButton® technology as an objective instrument to measure hot flash dynamics, the investigators will validate the technology in 12 perimenopausal women ages 45-60 y and BMI 18.5-40 kg/m2 who experience greater than or equal to 4 hot flashes per day. First, the investigators will validate the iButton® technology against self-report (subjective) hot flash incidence in a real world, ambulatory condition (via a hot flash journal). Next, the investigators will validate the iButton® technology during a controlled, laboratory-stimulated hot flash using a tube-lined suit that circulates warm water uniformly around the lower limbs (Med-EngTM). During the stimulated hot flash, the investigators will simultaneously measure core body temperature, skin blood flow, skin temperature, sweat rate, and heart rate alongside the iButton® to correlate (confirm) the observed thermoregulatory changes and further assess validity. To date, existing studies using iButtons® to assess changes in skin temperature have been conducted.

Each subject will undergo a two-phased screening to determine eligibility. Pre-enrollment measurements will include standard anthropometrics (weight, height), vital signs (blood pressure, heart rate), fasting blood draw, and questionnaires, as well as a 7-day hot flash journal that captures frequency and severity screening. Post-enrollment measurements will include simultaneous objective (via iButtons®) and subjective (via self-report journal) hot flash recordings (i.e., field testing), as well as a final laboratory visit will be conducted at Louisiana State University's School of Kinesiology and include body composition assessment, as well as the following assessments during a stimulated hot flash -- core temperature, skin blood flow, skin temperature, sweat rate, and heart rate.

ELIGIBILITY:
Inclusion Criteria:

* Healthy female
* Ages 45-60 y
* BMI between 18.5 kg/m2 and 40 kg/m2 (inclusive)
* Self-reported ≥4 hot flashes per day (for 4 out of the 7 days) (via 7-d hot flash journal)
* Meets both criteria for "peri-menopause (late phase)" classification: (1) experiences menopause-related symptoms (including hot flashes); (2) has hot gone 12 months in a row without a menstrual cycle; however, has sometimes more than 60 days between cycles.
* Medically cleared for participation by the Medical Investigator

Exclusion Criteria:

* Current smokers, or having smoked within the last 3 months
* History of diabetes (or other metabolic diseases)
* History of neurological disease
* History of cardiovascular disease
* Taking hormone replacement therapy, or other therapies/supplements designed to reduce severity of menopause symptoms (e.g., hot flashes)
* Pregnant, planning to become pregnant, or currently breastfeeding

Ages: 45 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Women in the late-phase of perimenopause with frequent hot flashes.
Study Population: Women who are in the late phase of perimenopause (based on the STRAW+10 criteria).
Sampling Method: Non-Probability Sample
Enrollment: 12 (Actual)
Dates: Start 2018-09-07 (Actual); Primary Completion 2022-09-19 (Actual); Study Completion 2022-09-19 (Actual)

PRIMARY OUTCOMES:
Skin temperature (via iButton®) | 2 hours
  Skin temperatures will be continually monitored at 2 sites: the sternum (chest) and forearm, using iButton® technology during a single hot flash that is stimulated at the laboratory visit.

SECONDARY OUTCOMES:
Skin temperature (via BIOPAC) | 2 hours
  Skin temperatures will be continually monitored at 5 sites: the mid-thigh, sternum (chest), forearm, mid-biceps, and scapula, during a single hot flash that is stimulated at the laboratory visit.
Skin blood flow (via laser-Doppler flowmetry) | 2 hours
  Skin blood flow will be measured continuously using a laser Doppler flowmeter on the sternum with the associated software (Perimed, Stockholm, Sweden) during a single hot flash that is stimulated at the laboratory visit.
Core temperature (via pill telemetry) | 2 hours
  Core temperature will be measured from an ingestible pill telemetry system (HTI Technologies; Palmetto, FL) during a single hot flash that is stimulated at the laboratory visit.
Sweat rate (via ventilated capsule) | 2 hours
  Sweat rates of the sternum and forearm will be measured using ventilated capsules secured with surgical adhesive during a single hot flash that is stimulated at the laboratory visit.

CONTACTS AND LOCATIONS:
Overall Officials: Kara L Marlatt, PhD, MPH, Principal Investigator — Pennington Biomedical Research Center
Locations (1):
- Pennington Biomedical Research Center, Baton Rouge, Louisiana, United States